CLINICAL TRIAL: NCT07391787
Title: Low-acid Contrast Media for Preventing Post ERCP Pancreatitis: a Multicenter, Retrospective, Cohort Study
Brief Title: Low-acid Contrast Media for Preventing Post ERCP Pancreatitis
Acronym: LAMP-R
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Professor of Medicine, Shandong University
Other Study IDs: KYLL-2025-12-013
Record Dates: First submitted 2026-01-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: Endoscopic retrograde cholangiopancreatography; Post ERCP pancreatitis; Contrast media; pH values
MeSH Terms: interventions — ioversol; iopromide; Iohexol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ioversol: Acidic contrast media, ioversol is used for radiography during ERCP procedure.
  Interventions: Drug: Ioversol
- Iopromide: Neutral contrast media, iopromide is used for contrast during ERCP procedure.
  Interventions: Drug: Iopromide
- Iohexol: Alkaline contrast media, iohexol is used for contrast during ERCP procedure.
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Ioversol — Ioversol was used for intervention in the ERCP procedure, while iopromide was used for controlled. ERCP was performed using endoscopes from different suppliers, and the guidewire assisted method were used for the papillary intubation.
  Groups: Ioversol
Drug: Iopromide — Iopromide was used for ERCP procedure as controlled group. ERCP was performed using endoscopes from different suppliers, and the guidewire assisted method were used for the papillary intubation.
  Groups: Iopromide
Drug: Iohexol — Iohexol was used for intervention in the ERCP procedure, while iopromide was used for controlled. ERCP was performed using endoscopes from different suppliers, and the guidewire assisted method were used for the papillary intubation.
  Groups: Iohexol

SUMMARY:
Title： Low-acid contrast media for preventing post ERCP pancreatitis: a multicenter, retrospective, cohort study (LAMP-R) .

Objective:

Main objective: This study aims to determine whether low-acid contrast media can reduce the incidence of post-ERCP pancreatitis.

Secondary objective: To investigate the severity of post-ERCP pancreatitis, the incidence rate of other complications, and the risk factors associated with different pH values of contrast media.

Research Design：Multicenter, retrospective cohort study.

Research participants:

Inclusion criteria: Patients aged 18 to 90 years who underwent ERCP diagnostic and therapeutic procedures were included consecutively.

Exclusion criteria: Patients who did not use contrast medium during ERCP, failed ERCP papillary intubation, developed acute pancreatitis within 3 days before surgery, ERCP stent removal/replacement, had a history of pancreaticoduodenectomy or biliary-enteric anastomosis, and whose postoperative amylase/lipase levels could not be traced were excluded.

Outcomes:

1. The rate of post-ERCP pancreatitis and severity of PEP 2. The rate of infection 3. The rate of gastrointestinal bleeding 4. The rate of perforation.

Sample size calculation:

A total of approximately 3,881 eligible ERCP patients were included from five tertiary Grade A centers. Specifically, 2,305 patients were from Qilu Hospital of Shandong University, 463 from Linyi People's Hospital, 121 from Qilu Third Hospital of Shandong University, 106 from Dezhou Hospital of Qilu Hospital of Shandong University, and 886 from Shengli Oilfield Central Hospital.

Statistical analysis SPSS 27 is used for statistics and analysis, including descriptive analysis, single-factor and multi-factor logistic regression analysis, analysis of variance, t-test, propensity score matching (PSM), etc. Categorical data are presented as counts and proportions, while continuous data are presented as mean ± standard deviation, depending on the distribution. Categorical data are analyzed using χ2 and Fisher's exact test, and continuous data are analyzed using Student's t-test or Mann-Whitney U test. Primary and secondary outcomes are presented as relative risks (RRs) with 95% confidence intervals (CIs).

DETAILED DESCRIPTION:
Introduction

1. The Clinical Burden of Post-ERCP Pancreatitis (PEP) Endoscopic Retrograde Cholangiopancreatography (ERCP) is a standard procedure for the diagnosis and treatment of pancreatobiliary diseases. However, it is associated with significant complications, among which post-ERCP pancreatitis (PEP) is the most frequent, occurring in 3-10% of all procedures and in 15-20% of high-risk patients. Despite continuous improvements in techniques and preventive strategies, PEP remains a major concern as it prolongs hospitalization, increases healthcare costs, and in severe cases, leads to substantial morbidity and mortality.
2. Contrast Media as a Potential Etiological Factor in PEP. The pathogenesis of PEP is multifactorial and not fully understood, involving mechanical, thermal, enzymatic, and chemical insults. A key procedural step in ERCP is the injection of contrast media into the pancreaticobiliary ducts. The resultant increase in hydrostatic pressure and the potential chemical irritation of the pancreatic ductal epithelium are hypothesized to trigger the inflammatory cascade leading to PEP. Emerging preclinical evidence suggests that the physicochemical properties of contrast media, particularly acidity (pH), may be a critical modifiable risk factor. Basic science studies indicate that low-pH contrast agents can exacerbate pancreatic injury through TRPV1-dependent pathways and by inducing abnormal calcium signaling, activating NF-κB and calcineurin pathways in acinar cells. For instance, injecting a contrast medium at pH 6.9 caused significant pancreatic edema and damage in animal models, while a solution at pH 7.3 caused minimal injury. These findings highlight a compelling biological plausibility for investigating contrast media characteristics in clinical PEP, yet high-quality clinical evidence is currently lacking.
3. Rationale and Focus of the Present Study. Building on the mechanistic hypothesis that acidity matters, we conducted preliminary measurements of three commonly used iso-osmolar non-ionic monomeric contrast agents (Iohexol, Iopromide, Ioversol). Notably, after 1:1 dilution with sterile water (a common practice in ERCP), the pH values differ: Iopromide (7.13~7.32), Ioversol (6.54~6.86), and Iohexol (7.25~7.46). This presents a natural experiment to evaluate whether these variations in acidity (pH) influence PEP risk in a real-world clinical setting.

Research method:

A multi-center, retrospective, cohort study.

Date collection:

From the HIS system, the following patient data will be collected: Demographics and History: Gender, age, clinical symptoms, whether it is the first ERCP procedure, history of previous PEP, history of Sphincter of Oddi Dysfunction (SOD). Laboratory Tests (pre- and post-ERCP): White blood cell count, hemoglobin, C-reactive protein, procalcitonin, ALT, AST, GGT, ALP, total bilirubin, direct bilirubin, amylase, lipase. Imaging Studies: CT, EUS, MRCP findings. Medication & Procedural Details (from order sheets): Type of contrast media used during ERCP, perioperative use of rectal NSAIDs (e.g., indomethacin suppository), postoperative antibiotic use (yes/no and specific agents). Post-Operative Clinical Course (from medical and nursing records): Occurrence of new abdominal pain (with NRS score), fever (maximum temperature and duration), hematemesis or melena. For PEP patients: length of prolonged hospitalization, severity of PEP (graded based on extended hospital stay and imaging findings).

From the Endoscopic Quality Control System, the following procedural details will be collected: Papillary Anatomy & Cannulation: Peri-diverticular papilla, difficult cannulation, guidewire entry into the pancreatic duct. Performance of pancreatography, visualization of side branches, pancreatobiliary ductal anomalies. Pre-cut sphincterotomy, papillary balloon dilation (standard or large-balloon), endoscopic sphincterotomy (EST) with size classification (small, medium, large). Biliary Disease Specifics (if applicable): Common bile duct (CBD) diameter (<1.0 cm), presence of CBD stones, stone size (<1.0 cm), stone extraction method (balloon vs. basket), placement of a pancreatic duct stent. Final diagnosis, total procedure duration. Stricture Characterization (if applicable): Pathological classification of any stricture (benign, malignant, indeterminate).

Research protocol:

1. This study retrospectively collected endoscopic retrograde cholangiopancreatography (ERCP) diagnosis and treatment data from five tertiary hospitals. Including patient's information, ERCP procedurel details, and postoperative adverse events were documented in a standardized record form. Data from each participating center were first desensitized and corrected by local data quality control personnel before being consolidated at the main center. The ERCP quality control administrator of the research center then performed unified data desensitization and homogenization to ensure information security and reliable data quality.
2. Based on the type of contrast agent used during ERCP, patients were categorized into three groups: the acidic contrast agent group (Ioversol), the neutral contrast agent group (Iopromide), and the alkaline contrast agent group (Iohexol). An overall assessment of the data was conducted, and univariate and multivariate Logistic regression analyses were performed to identify high-risk factors for post-ERCP pancreatitis (PEP). Both study-derived and well-established PEP risk factors were included as covariates. Using the neutral contrast agent group as the control, propensity score matching (PSM) was applied to match ERCP data from the acidic and alkaline contrast agent groups with the neutral contrast agent group, resulting in two separate matched datasets: acid vs. neutral contrast agent and alkaline vs. neutral contrast agent. Balance testing was performed on both matched sets to ensure standardized differences were below 10%, confirming the appropriate the matching.
3. Finally, two-sample chi-square tests were used to compare the incidence of PEP between the acidic and neutral contrast agent groups and between the alkaline and neutral contrast agent groups, investigating the influence of contrast agent acidity on PEP in a real-world setting.

Outcomes： Primary outcome: The rate of post-ERCP pancreatitis: According to the Cotton criteria and consensus opinions, postoperative pancreatitis is defined as new-onset upper abdominal pain after surgery, with amylase or lipase levels elevated to three times the upper limit of normal, and an extended hospital stay of at least 2 nights.

Secondary outcomes: The severity of post-ERCP pancreatitis and other post-ERCP complications. The severity of PEP is defined as follows: mild pancreatitis requires an extended hospital stay of 2 to 3 days, moderate pancreatitis requires an extended hospital stay of 4 to 10 days, and severe pancreatitis requires an extended hospital stay of more than 10 days. The rate of infection: Postoperative fever (Tmax > 38°C, >24 hours, and excluding infections in other sites, such as pulmonary infection, urinary tract infection, etc.); WBC > 10*10^9/L or < 3*10^9/L, with elevated infection indicators (elevated CRP, PCT); imaging findings suggestive of cholangitis, peribiliary effusion, etc. The rate of bleeding: Postoperative hematemesis or black stool; postoperative hemoglobin (HGB) decrease of more than 20g/L compared to preoperative levels, or requiring blood transfusion; postoperative changes in vital signs (such as increased heart rate, decreased blood pressure, pale complexion, etc.); postoperative emergency endoscopic exploration for hemostasis or imaging findings indicating bleeding in the biliary-pancreatic system, or requiring emergency DSA treatment. The rate of perforation: Postoperative abdominal pain emerges, imaging reveals gas accumulation around the biliary-pancreatic region, or ERCP suggests a potential perforation.

Definition:

Difficult intubation: The surgical record describes it as difficult intubation, with the guidewire repeatedly entering the pancreatic duct. Double guidewire-assisted intubation or pre-cut sphincterotomy-assisted intubation was performed.

Branch pancreatic duct visualization: Defined as the clear visualization of the branch pancreatic duct in ERCP images, or the surgical record describing the presence of visible branch pancreatic duct.

Anatomic abnormalities of the pancreaticobiliary duct: including pancreas divisum, abnormal pancreaticobiliary junction, annular pancreas, and congenital choledochal cyst.

Trans-papillary precut: including trans-pancreaticobiliary sphincter precut, trans-papillary needle knife precut, and fenestration.

EPLBD: A lagre balloon with a diameter of ≥12mm is used to dilate the Oddi's sphincter.

Nipple incision size: Small incision is defined as an incision smaller than 1/3 of the distance from the nipple opening to the lateral edge of the mouth. Medium incision is defined as an incision larger than 1/3 but smaller than 1/2 of this distance. Large incision is defined as an incision larger than 2/3 of this distance.

Operation duration: Defined as the time from the start of nipple cannulation to the end of the operation, representing the time difference between the nipple imaging time and the X-ray time for stent or biliary drainage tube placement in the system workstation.

ERCP failure: defined as failure of papillary cannulation, with no contrast medium injected into the biliary-pancreatic duct.

Quality Control:

To ensure data consistency and quality, data collection is supervised by the principal investigator at each center. All data are then sent to the main center for centralized statistical verification and analysis.

Research plan： August, 2025 - June, 2026.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years who underwent ERCP diagnostic and therapeutic procedures were included consecutively.

Exclusion Criteria:

* Patients who did not use contrast media during ERCP
* Failed ERCP papillary intubation
* Patients with acute pancreatitis within 3 days before ERCP
* ERCP stent removal/replacement
* Patients who had a history of pancreaticoduodenectomy or biliary-enteric anastomosis
* Patients whose postoperative amylase/lipase levels could not be traced.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of approximately 3,881 eligible ERCP patients were included from five tertiary Grade A centers. All patients signed the informed consent form. Specifically, 2,305 patients were from Qilu Hospital of Shandong University, 463 from Linyi People's Hospital, 121 from Qilu Third Hospital of Shandong University, 106 from Dezhou Hospital of Qilu Hospital of Shandong University, and 886 from Shengli Oilfield Central Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3979 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
The rate of Post-ERCP pancreatitis | Assessed up to 3 days after ERCP procedure.
  According to the Cotton criteria and consensus opinions, post-ERCP pancreatitis is defined as new-onset upper abdominal pain after surgery, with amylase or lipase levels elevated to three times the upper limit of normal, and an extended hospital stay of at least 2 nights.

SECONDARY OUTCOMES:
The severity of post-ERCP pancreatitis | Assessed up to 10 days after ERCP procedure.
  The severity of PEP is defined as follows: mild pancreatitis requires an extended hospital stay of 2 to 3 days, moderate pancreatitis requires an extended hospital stay of 4 to 10 days, and severe pancreatitis requires an extended hospital stay of more than 10 days.
The rate of infection | Assessed up to 3 days after ERCP procedure.
  Postoperative fever (Tmax > 38°C, >24 hours, and excluding infections in other sites, such as pulmonary infection, urinary tract infection, etc.); WBC > 10*10^9/L or < 3*10^9/L, with elevated infection indicators (elevated CRP, PCT); imaging findings suggestive of cholangitis, peribiliary effusion, etc.
The rate of gastrointestinal bleeding | Assessed up to 3 days after ERCP procedure.
  Gastrointestinal bleeding: Postoperative hematemesis or black stool; postoperative hemoglobin (HGB) decrease of more than 20g/L compared to preoperative levels, or requiring blood transfusion; postoperative changes in vital signs (such as increased heart rate, decreased blood pressure, pale complexion, etc.); postoperative emergency endoscopic exploration for hemostasis or imaging findings indicating bleeding in the biliary-pancreatic system, or requiring emergency DSA treatment.
Perforation | Assessed up to 3 days after ERCP procedure.
  Perforation: Postoperative abdominal pain emerges, imaging reveals gas accumulation around the biliary-pancreatic region, or ERCP suggests a potential perforation.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong
  - Qilu hospital, Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No